CLINICAL TRIAL: NCT04272307
Title: MIcroorganisms as Triggers in Acute Severe Ulcerative Colitis and Their Influence on Medical Therapy Efficacy: a Multi-omics Pilot Approach.
Acronym: ITAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/28
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases; Colitis; Ulcerative
Keywords: Inflammatory Bowel Disease; Acute severe ulcerative colitis; Microbiome; Prognostic factors
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis; Ulcer | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample, stool and colonic biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Severe Ulcerative Colitis group
  Interventions: Biological: Blood samples; Procedure: Stool samples; Procedure: Colorectal biopsies
- Non-severe Ulcerative Colitis group
  Interventions: Biological: Blood samples; Procedure: Stool samples; Procedure: Colorectal biopsies

INTERVENTIONS:
Biological: Blood samples — At inclusion, at day 5, day 42 and at 3 months, one 2 ml EDTA blood tube will be collected for metabolomics.
  Polar metabolites, lipids, free fatty acids and bile acids will be identified and quantitated using ultra high-performance liquid chromatography/tandem accurate mass spectrometry method.
  At inclusion, one 2 ml EDTA tube will be stored as a DNA collection.
Procedure: Stool samples — One stool sample will be taken at baseline, day 5, day 42 and at 3 months and frozen at -80°C and divided in 2 aliquots.
  One stool aliquot will be used for metabolomics. Polar metabolites, lipids, free fatty acids and bile acids will be identified and quantitated using ultra high-performance liquid chromatography/tandem accurate mass spectrometry method. The other one will be used for microbiota analysis. Samples will be sent to the McGill University (Prof. SALEH's lab) for extraction and then, Génome Québec Innovation Centre (McGill University, Montréal, Canada) for sequencing of the V4 region of the 16S rRNA gene on Illumina MiSeq in paired-end mode.
Procedure: Colorectal biopsies — During routine flexible sigmoidoscopy, 6 biopsies will be collected with a 5 mm biopsy forceps at baseline and at 3 months. Biopsies will be placed into a sterile vial containing RNAlater (Qiagen, Hilden, Germany) and stored at -80°C. Two biopsies will be used for mucosal microbiome analysis in the same way as the stool sample. Four biopsies will be used for RNAseq. Samples will be shipped to Prof. SALEH's lab in Montréal for nucleic acid extraction. The McGill University and Génome Québec Innovation Centre (McGill University, Montréal, Canada) will provide library preparation and next generation sequencing. The average number of uniquely mapped reads per sequencing run will be 30 million reads per sample.

SUMMARY:
This pilot prospective study will investigate the role of microbiota and known enteropathogens in Acute Severe Ulcerative Colitis (ASUC). Investigators will compare a group of patients hospitalized for an ASUC with patients experiencing a Non-Severe Ulcerative Colitis (NSUC) flare by investigating microbiome, metabolome and transcriptome and integrating this data through a multi-omic framework. This systems biology approach aims at enhance our understanding of this severe event, define diagnosis and prognosis biomarkers to improve medical therapy and avoid colectomy and/or death.

DETAILED DESCRIPTION:
Ulcerative Colitis (UC) is one of the two entities of Inflammatory Bowel Disease (IBD), along with Crohn's disease. One in 4 patients experiences an Acute Severe Ulcerative Colitis (ASUC) during the disease course, defined as a severe flare with systemic inflammation. ASUC is a medical and surgical emergency as complications and death may occur when patients do not respond to medical therapy and require salvage colectomy. Little is known about the pathophysiology and specifically the triggers of ASUC. At baseline, investigators will investigate the presence of a microbiome signature in patients with an ASUC compared with patients with a non-severe UC flare (NSUC). To identify the role of microorganisms, investigators will look specifically for known enteropathogens, i.e. Clostridium difficile and Cytomegalovirus. Investigators will investigate the impact of microbiota disruptors, such as antibiotics, NSAIDs and diet on microbiota and patients' outcomes. To evaluate the role of the host inflammatory pathways, investigators will study the colonic mucosa transcriptome and the host metabolome, focusing on anti-microbial defence pathways, regarding the suggested role of defective immune defence pathways in IBD pathogenesis. Investigators will focus on the IL23 and Jak pathways, since new drugs targeting these molecules are now available for IBD patients but still not recommended in the ASUC setting. Our last approach will be to evaluate the predictability of the response to therapy according to baseline and early changes of stool microbiome and host metabolome.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Adult patients diagnosed with Ulcerative Colitis according to usual criteria.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

ASUC group:

Adult patients hospitalized an ASUC defined according to Truelove criteria, i.e. ≥6 bloody daily stools with one or more of the following criteria: temperature >37.8°C, pulse >90 beats/min, haemoglobin <10.5g/dl or C Reactive-Protein >45mg/l.

Non severe acute UC patients (NSUC) group:

Adult patients with disease activity symptoms, corresponding to a partial Mayo score of 4 or more with a rectal bleeding subscore of at least 1, without Truelove severity criteria.

Exclusion Criteria:

* Patients with perianal lesions, ileal lesions or endoscopic aspect of the colonic lesions related to a Crohn's disease acute severe colitis.
* Patients under 18 years old.
* Patients under legal protection or unable to express their consent.
* Patients not affiliated to a health insurance system.
* Patients deprived of liberty by judiciary or administrative decision or hospitalized without consent or admitted in a sanitary or social institution for another reason than research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Ulcerative Colitis according to usual criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Analysis of the faecal microbiota in each group. | Inclusion Visit
  Sequencing of the V4 region of the 16S rRNA gene at inclusion on the colonic biopsies taken during routine sigmoidoscopy.

SECONDARY OUTCOMES:
Diagnosis of Clostridium difficile infections | Inclusion Visit
  Investigators will define a Clostridium difficile infection as Glutamate dehydrogenase positive test associated to Polymerase Chain Reaction Toxin positive test in the stool or intestinal fluid.
Diagnosis of Cytomegalovirus (CMV) infections | baseline
  Investigators will define a CMV infection as presence of CMV inclusions in Hemalum Eosine or ImmunoHistoChemistry in the colonic biopsies taken during the baseline sigmoidoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No